CLINICAL TRIAL: NCT04622904
Title: The Effect of Intravenous Infusions of Lidocaine and Magnesium Versus Lidocaine and Ketamine Versus Lidocaine Alone on Recovery Profile and Postoperative Pain After Elective Gynecological Surgery
Brief Title: Lidocaine and Magnesium and Ketamine in Gynecological Surgery
Acronym: annie-sophia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 11/2020
Record Dates: First submitted 2020-10-31; First posted 2020-11-10 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Pain, Postoperative; Pain, Acute; Pain, Chronic; Pain, Neuropathic; Lidocaine; Ketamine; Magnesium; Central Nervous System Depressants; Analgesics; Neurotransmitter Agents; Analgesics, Non-narcotic
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Chronic Pain; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lidocaine-magnesium group (Active Comparator): combination of lidocaine and magnesium infusions
  Interventions: Drug: lidocaine-magnesium infusion
- lidocaine-ketamine group (Active Comparator): combination of lidocaine and ketamine infusions
  Interventions: Drug: lidocaine-ketamine infusion
- lidocaine group (Active Comparator): lidocaine infusion alone
  Interventions: Drug: lidocaine infusion

INTERVENTIONS:
Drug: lidocaine-magnesium infusion — A bolus dose of lidocaine of 1.5 mg/kg will be administered within 10 minutes preoperatively diluted in 100 mL of saline. Then, 3 mg/kg/h of lidocaine will be administered intraoperatively. A bolus dose of ketamine of 0.35 mg/kg will be administered within 10 minutes preoperatively diluted in 100 mL of saline. Followingly, 0.2 mg/kg/h of ketamine will be administered intraoperatively diluted in a 60 mL syringe and administered at a rate of 20 mL/h
  Arms: lidocaine-magnesium group
Drug: lidocaine-ketamine infusion — A bolus dose of lidocaine of 1.5 mg/kg will be administered within 10 minutes preoperatively diluted in 100 mL of saline. Then, 3 mg/kg/h of lidocaine will be administered intraoperatively. A bolus dose of magnesium of 50 mg/kg will be administered within 10 minutes preoperatively diluted in 100 mL of saline. Followingly, 10 mg/kg/h of magnesium will be administered intraoperatively diluted in a 60 mL syringe and administered at a rate of 20 mL/h
  Arms: lidocaine-ketamine group
Drug: lidocaine infusion — A bolus dose of lidocaine of 1.5 mg/kg will be administered within 10 minutes preoperatively diluted in 100 mL of saline. Then, 3 mg/kg/h of lidocaine will be administered intraoperatively. A bolus dose of normal saline 100 mL will be administered preoperatively within 10 minutes. Followingly, normal saline will be administered intraoperatively at a rate of 20 mL/h
  Arms: lidocaine group

SUMMARY:
The aim of this study will be to investigate the effect of a combination of intravenous infusions of lidocaine and magnesium versus a combination of intravenous infusions of lidocaine and ketamine versus an intravenous infusion of lidocaine alone on recovery profile, quality of recovery and postoperative pain after elective gynecological surgery

DETAILED DESCRIPTION:
Inadequately treated postoperative pain after gynecological surgery may untowardly affect early recovery and also lead to the development of chronic pain. Opioid-based analgesia is associated with side-effects, such as respiratory depression, postoperative nausea and vomiting and occasional induction of tolerance and hyperalgesia. Therefore, in recent years research has focused on the quest for non-opioid-based regimens for perioperative analgesia in the context of multimodal analgesic techniques. These techniques have been shown to possess significant advantages, such as allowing earlier mobilization after surgery, early resumption of enteral feeding and reduced hospital length of stay.

In this context, the intraoperative intravenous injection of lidocaine has been reported to improve postoperative pain control, reduce opioid consumption and improve the quality of postoperative functional recovery after general anesthesia. Intraoperative infusions of ketamine (an N-methyl-D-aspartate receptor inhibitor) have also been correlated with reduced pain scores and a decrease in analgesic requirements postoperatively. Lastly, magnesium (acting through modification of the action of N-methyl-D-aspartate receptors) is another agent, which, as an adjuvant to general anesthesia may improve postoperative recovery and pain control through inhibition of cardiovascular response, reduction in general anesthetic needs, enhanced analgesia and anti-inflammatory response.

There is insufficient data in literature investigating the effect of combinations of these agents intraoperatively. It would be of interest to demonstrate whether the administration of combinations of infusions can lead to enhanced postoperative recovery, an improved opioid-sparing effect and a decrease in the development of chronic pain as compared to the administration of a sole agent alone. Therefore, the aim of this study will be to investigate the effect of a combination of intravenous infusions of lidocaine and magnesium versus a combination of intravenous infusions of lidocaine and ketamine versus an intravenous infusion of lidocaine alone on recovery profile, quality of recovery and postoperative pain after elective gynecological surgery.

ELIGIBILITY:
Inclusion Criteria:

* adult female patients
* American Society of Anesthesiologists (ASA) classification I-II
* elective open gynecological surgery

Exclusion Criteria:

* body mass index (BMI) >35 kg/m2
* contraindications to local anesthetic administration or non-steroidal agents administration
* systematic use of analgesic agents preoperatively
* chronic pain syndromes preoperatively
* neurological or psychiatric disease on treatment
* pregnancy
* severe hepatic or renal disease
* history of cardiovascular diseases/ arrhythmias/ conduction abnormalities
* drug or alcohol abuse
* language or communication barriers
* lack of informed consent

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only female patients are subjected to gynecological suregry
Enrollment: 90 (Estimated)
Dates: Start 2020-11-14 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
change from baseline in Quality of Recovery (QoR)-15 score after surgery | 24 hours postoperatively
  The QoR-15 is a quality of recovery scale that consists of 15 questions (items),including questions regarding pain (2 items), physical comfort (5 items), self-care ability (2 items), psychological support (2 items) and emotional state (4 items). Every item is scored on a scale of 10, with the lowest total score of 0 and the highest score of 150. The higher the score, the better the recovery quality of the patient
pain score on arrival to Post-Anesthesia Care Unit (PACU) | immediately postoperatively
  pain score by the use of Numeric Rating Scale (NRS) on arrival to PACU, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score at discharge from Post-Anesthesia Care Unit (PACU) | at discharge from PACU, approximately 1 h postoperatively
  pain score by the use of Numeric Rating Scale (NRS) at discharge from PACU, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 3 hours postoperatively | 3 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 3 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 6 hours postoperatively | 6 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 6 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 24 hours postoperatively | 24 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 24 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 48 hours postoperatively | 48 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 48 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"

SECONDARY OUTCOMES:
Post Anesthesia Care Unit (PACU) duration of stay | immediately postoperatively
  duration of patient stay at PACU
sedation on arrival to Post-Anesthesia Care Unit | immediately postoperatively
  sedation will be assessed with a 5-point sedation scale, where: 1, patient perfectly conscious; 2, patient feels a little drowsy; 3, patient seems to be sleeping but immediately reacts to verbal stimulation; 4, patient seems to be sleeping but slowly reacts to verbal stimulation and 5, patient seems to be sleeping and does not react to verbal stimulation but does react to a stimulus such as shaking or pain
sedation at discharge from Post-Anesthesia Care (PACU) Unit | at discharge from PACU, approximately 1 hour postoperatively
  sedation will be assessed with a 5-point sedation scale, where: 1, patient perfectly conscious; 2, patient feels a little drowsy; 3, patient seems to be sleeping but immediately reacts to verbal stimulation; 4, patient seems to be sleeping but slowly reacts to verbal stimulation and 5, patient seems to be sleeping and does not react to verbal stimulation but does react to a stimulus such as shaking or pain
sevoflurane consumption during general anesthesia | change of sevoflurane vaporizer weight from before induction to end of anesthesia, an average period of 2 hours
  the sevoflurane vaporizer will be weighed before anesthetic induction and at the end of anesthesia and consequently sevoflurane consumption during anesthesia will be determined
time to first request for analgesia | during stay in Post-Anesthesia Care Unit, approximately 1 hour postoperatively
  the time for the first patient request for analgesia will be noted
morphine consumption in Post-Anesthesia Care Unit (PACU) | immediately postoperatively
  mg of morphine requested during patient PACU stay
morphine consumption in the first 48 hours | 48 hours postoperatively
  patients will be followed for cumulative morphine consumption through patient-controlled analgesia device for 48 hours postoperatively
sleep quality | 24 hours postoperatively
  subjective evaluation of sleep quality by patients, based on a sleep questionnaire (evaluation of sleep duration, number of nocturnal awakenings and marking of sleep quality)
first mobilization after surgery | 24 hours postoperatively
  patients will be questioned regarding the time at which they mobilized after surgery
gastrointestinal recovery after surgery | 48 hours postoperatively
  patients will be questioned regarding the time they first felt enteral sounds and the time they had their first flatus after surgery
satisfaction from postoperative analgesia | 24 hours postoperatively
  satisfaction from postoperative analgesia on a six-point Likert scale with 1 marked as minimal satisfaction and 6 as maximal satisfaction
first fluid intake | 48 hours postoperatively
  patients will be questioned regarding the time they had their first fluid intake
first solid intake | 48 hours postoperatively
  patients will be questioned regarding the time they had their first solid intake
hospitalization time | 96 hours postoperatively
  duration of hospital stay after surgery in days
fentanyl requirement during surgery | intraoperatively
  dose of required fentanyl intraoperatively to maintain systolic arterial blood pressure and heart rate within the 20% of baseline value
side effects intraoperatively | intraoperatively
  patients will be monitored for side-effects of the administered agents intraoperatively
side effects postoperatively | 72 hours postoperatively
  patients will be monitored for side-effects of the administered agents postoperatively
incidence of chronic pain 1 month after surgery | 1 month after surgery
  occurrence of chronic pain at the site of the operation 1 month after surgery, with the use of the Numeric Rating Scale (NRS), at rest and during movement
incidence of chronic pain 3 months after surgery | 3 months after surgery
  occurrence of chronic pain at the site of the operation 3 months after surgery, with the use of the Numeric Rating Scale (NRS), at rest and during movement

OTHER OUTCOMES:
time to emergence | end of operation, approximately 2 hours after start of surgery
  time from sevoflurane discontinuation to first patient response (eye opening)
time to extubation | end of operation, approximately 2 hours after start of surgery
  time from sevoflurane discontinuation to tracheal extubation

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, DESA, Principal Investigator — Aretaieion University Hospital
Locations (1):
- Aretaieion University Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brandsborg B, Nikolajsen L. Chronic pain after hysterectomy. Curr Opin Anaesthesiol. 2018 Jun;31(3):268-273. doi: 10.1097/ACO.0000000000000586. PMID 29474214
- [Background] Helander EM, Webb MP, Bias M, Whang EE, Kaye AD, Urman RD. Use of Regional Anesthesia Techniques: Analysis of Institutional Enhanced Recovery After Surgery Protocols for Colorectal Surgery. J Laparoendosc Adv Surg Tech A. 2017 Sep;27(9):898-902. doi: 10.1089/lap.2017.0339. Epub 2017 Jul 25. PMID 28742434
- [Background] Herroeder S, Pecher S, Schonherr ME, Kaulitz G, Hahnenkamp K, Friess H, Bottiger BW, Bauer H, Dijkgraaf MG, Durieux ME, Hollmann MW. Systemic lidocaine shortens length of hospital stay after colorectal surgery: a double-blinded, randomized, placebo-controlled trial. Ann Surg. 2007 Aug;246(2):192-200. doi: 10.1097/SLA.0b013e31805dac11. PMID 17667496
- [Background] Sen H, Sizlan A, Yanarates O, Emirkadi H, Ozkan S, Dagli G, Turan A. A comparison of gabapentin and ketamine in acute and chronic pain after hysterectomy. Anesth Analg. 2009 Nov;109(5):1645-50. doi: 10.1213/ANE.0b013e3181b65ea0. PMID 19843803
- [Background] Haryalchi K, Abedinzade M, Khanaki K, Mansour Ghanaie M, Mohammad Zadeh F. Whether preventive low dose magnesium sulphate infusion has an influence on postoperative pain perception and the level of serum beta-endorphin throughout the total abdominal hysterectomy. Rev Esp Anestesiol Reanim. 2017 Aug-Sep;64(7):384-390. doi: 10.1016/j.redar.2016.11.009. Epub 2017 Feb 14. English, Spanish. PMID 28214095
- [Background] Xu SQ, Li YH, Wang SB, Hu SH, Ju X, Xiao JB. Effects of intravenous lidocaine, dexmedetomidine and their combination on postoperative pain and bowel function recovery after abdominal hysterectomy. Minerva Anestesiol. 2017 Jul;83(7):685-694. doi: 10.23736/S0375-9393.16.11472-5. Epub 2017 Jan 17. PMID 28094477
- [Background] Garcia-Navia JT, Tornero Lopez J, Egea-Guerrero JJ, Vilches Arenas A, Vazquez Gutierrez T. Effect of a single dose of lidocaine and ketamine on intraoperative opioids requirements in patients undergoing elective gynecological laparotomies under general anesthesia. A randomized, placebo controlled pilot study. Farm Hosp. 2016 Jan 1;40(1):44-51. doi: 10.7399/fh.2016.40.1.9339. PMID 26882833
- [Background] Arikan M, Aslan B, Arikan O, Horasanli E, But A. Comparison of the effects of magnesium and ketamine on postoperative pain and morphine consumption. A double-blind randomized controlled clinical study. Acta Cir Bras. 2016 Jan;31(1):67-73. doi: 10.1590/S0102-865020160010000010. PMID 26840358